CLINICAL TRIAL: NCT05488132
Title: Application of Anti-siglec-6 CAR-T Cell Therapy in Relapsed and Refractory Acute Myeloid Leukemia (rr/AML)
Brief Title: Administration of Anti-siglec-6 CAR-T Cell Therapy in Relapsed and Refractory Acute Myeloid Leukemia (rr/AML)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, President, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2022-KL119-01
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia Refractory; Acute Myeloid Leukemia, in Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-siglec-6 CAR-T cell therapy (Experimental): anti-siglec-6 CAR-T cell therapy
  Interventions: Drug: anti-siglec-6 CAR-T cell therapy

INTERVENTIONS:
Drug: anti-siglec-6 CAR-T cell therapy — Enrolled patients will receive prespecified dose of autologous CAR-T cells.

SUMMARY:
To evaluate the safety and efficacy of anti-Siglec-6 CAR-T cells in the treatment of relapsed and refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
Sialic acid-binding immunoglobulin-like lectins (Siglec) are a class of classical immunoglobulin-like lectins. Studies have shown that Siglec-6 is commonly expressed in AML but not detected on normal hematopoietic stem and progenitor cells (HSC/P). In vitro experiments revealed that anti-Siglec-6 CAR-T cell treatment did not affect the viability or lineage differentiation in colony-forming assays. These data suggest that anti-SigLlec-6 is an ideal target with great potential for treating acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must sign and date the Informed Consent before initiating any study specific procedures or activities;
2. At the age of 18-70 years old;
3. Diagnosed as relapse/refractory (r/r) de novo or secondary acute myeloid leukemia (AML);
4. The patient has recovered from the toxicity of previous treatment;
5. ECOG score ≤ 2 and expected survival period is not less than 3 months;
6. Adequate organ function defined as:AST ≤3×ULN; ALT ≤3×ULN; Total bilirubin ≤1.5×ULN; Serum creatinine ≤1.5×ULN, or CCR≥60 mL/min; Hemoglobin ≥60g/L ; Indoor oxygen saturation ≥92%; LVEF≥45%;
7. Pregnancy testing: females of childbearing potential must have a negative serum or urine pregnancy test;
8. From the use of study drug to 2 years after treatment, males and female of childbearing potential must agree to use an effective method of contraception.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia;
2. History or presence of a CNS disorder;
3. HBsAg is positive; HCV 、HIV or Syphilis antibody are positive, CMV DNA in peripheral blood is more than≥500 copies /mL;
4. History of severe hypersensitivity reaction;
5. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, atrial fibrillation, or other clinically significant cardiac disease within 12 months before enrollment;
6. History of organ transplant surgery;
7. Required systemic application of immunosuppressive or other drugs;
8. Auto-SCT within the 3 months before enrollment;
9. Active autoimmune or inflammatory diseases of the nervous system (e.g., Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically active cerebrovascular diseases (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES));
10. Requirement for urgent therapy due to ongoing or impending oncologic emergency (eg, leukostasis or tumor lysis syndrome (TLS)) ;
11. Presence or suspicion of a fungal, bacterial, viral, or other infection that is uncontrolled or requiring antimicrobials for management;
12. Live vaccine received within the ≤ 4 weeks before enrollment;
13. Persons with serious mental illness;
14. History of major surgical operations four weeks before enrollment;
15. History of alcoholism or substance abuse;
16. Was identified by the investigators as unsuitable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | Baseline up to 28 days after T cell infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
MRD negative overall response rate (MRD- ORR) | 3 months
  Assessment of MRD negative overall response rate (MRD- ORR) at 3 months of treatment
Overall response rate (ORR) | Month 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi ) at Month 6, 12, 18 and 24
Event-free survival (EFS) | Month 6, 12, 18 and 24
  Assessment of EFS at Month 6, 12, 18 and 24
Overall survival (OS) | Time Frame: Month 6, 12, 18 and 24
  Assessment of OS at Month 6, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, M.D., Ph.D., Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- Kailin Xu, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No